CLINICAL TRIAL: NCT06641037
Title: A Phase 1, Open-label, Randomized, Crossover Study to Assess the Effect of Food on the Pharmacokinetics of LY3866288 in Healthy Participants
Brief Title: A Study of LY3866288 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27311; J4G-OX-JZVC (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3866288 Cohort 1 (High-Fat Meal) (Experimental): LY3866288 single and multiple capsules administered orally under fasted/fed conditions in cross-over manner within cohort
  Interventions: Drug: LY3866288
- LY3866288 Cohort 2 (Low-Fat Meal) (Experimental): LY3866288 single and multiple capsules administered orally under fasted/fed conditions in cross-over manner within cohort
  Interventions: Drug: LY3866288

INTERVENTIONS:
Drug: LY3866288 — Administered orally

SUMMARY:
The purpose of this study is to evaluate how well LY3866288 is tolerated and what side effects may occur in healthy participants. The study drug will be administered orally. Blood tests will be performed to check how much LY3866288 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 9 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Females must be of nonchildbearing potential or of childbearing potential and agree to use contraception
* Males must either be infertile via bilateral orchiectomy or vasectomized at least 90 days prior to screening with proper documentation
* Body mass index (BMI) between 18.5 and 32.0 kilogram per square meter (kg/m²)
* In good general health, determined by no clinically significant findings from medical history, physical examination, 12 lead electrocardiogram (ECGs), vital signs measurements, or clinical laboratory evaluations at screening and/or check-in as assessed by the investigator (or designee)

Exclusion Criteria:

* Females only: Are lactating or pregnant
* Any history or presence of disease(s), deemed clinically significant:

  * Dermatological disease
  * Liver disease
  * Metabolic disease, including congenital nonhemolytic hyperbilirubinemia (e.g., Gilbert syndrome)
  * Gastrointestinal disease, including peptic ulcer disease, active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the study drug, or gastric reduction surgery. Note: participants with a history of appendectomy and/or inguinal hernia repairs will be acceptable
  * Biliary disease, including cholecystectomy
  * Cancer within the past 5 years (except localized basal cell, squamous, or in situ cancer of the skin)
  * History or current evidence of ophthalmic disorder, such as central serous retinopathy or retinal vein occlusion, active wet age-related macular degeneration, diabetic retinopathy with macular edema, uncontrolled glaucoma, corneal pathology such as keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration
  * Clinically significant, active cardiovascular disease or history of myocardial infarction within 6 months prior to first dose, or 12-lead ECG abnormalities that are clinically significant at screening
* History of alcohol and/or drug abuse within 2 years prior to screening
* Have been on a diet incompatible with the on-study diet, in the opinion of the investigator (or designee), and as confirmed by the sponsor, within the 30 days prior to Day 1 and throughout
* Use of tobacco, smoking cessation products, products containing nicotine, or e-cigarettes (nicotine and non-nicotine) within 90 days prior to screening and throughout

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration of LY3866288 | Baseline to Study Completion (Up to 3 Weeks)
  PK: AUC From Time 0 to the Time of the Last Quantifiable Concentration of LY3866288
PK: AUC Extrapolated to Infinity of LY3866288 | Baseline to Study Completion (Up to 3 Weeks)
  PK: AUC Extrapolated to Infinity of LY3866288
PK: Maximum Concentration (Cmax) of LY3866288 | Baseline to Study Completion (Up to 3 Weeks)
  PK: Cmax of LY3866288

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No